CLINICAL TRIAL: NCT04984642
Title: Plasma, Urine and Tear Omics Changes Based on Protein and Metabonomics Technology in Different Diets and Screening of Healthy Diet Markers
Brief Title: Plasma, Urine and Tear Omics Changes in Different Diets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2020-865
Record Dates: First submitted 2021-07-08; First posted 2021-07-30 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Diet, Healthy
MeSH Terms: interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- healty subject (Experimental)
  Interventions: Other: diet

INTERVENTIONS:
Other: diet — have OGTT,normal diet, high fat diet, low calorie diet, and ketogenic diet in turn

SUMMARY:
The study plans to start in July 2021, and it is expected that 20 healthy people (aged 18-70 years old, BMI 18.5-40kg/m2) will carry out a 5-week intervention and follow-up. Participants will be enrolled in the group through the screening and plan to take regular diet, OGTT, high-fat diet, low-calorie diet and ketogenic diet within 5 weeks. The proteomics and metabolomics indicators of tear, plasma, and urine specimens will be measured at 5 time points at baseline, 30 minutes, 1 hour, 2 hours, and 3 hours for each diet. The correlation of proteomics and metabolomics indicators with classic laboratory parameters (BMI, HDL, LDL, cholesterol, triglyceride levels, and insulin resistance (HOMA-IR)) will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy individuals aged 20-70 years, with a body mass index (BMI) of 18.5-40 kg/m².
2. No known chronic medical conditions.
3. Willingness to comply with study requirements and adhere to the intervention protocol.

Exclusion Criteria:

1. Presence of significant medical conditions or chronic diseases.
2. Diagnosis of diabetes mellitus or prediabetes.
3. Triglyceride level ≥4 mmol/L.
4. Blood pressure ≥160/100 mmHg or presence of malignant hypertension.
5. History of an eating disorder.
6. Previous bariatric surgery.
7. Severe gastrointestinal diseases.
8. History of diarrhea within the past two weeks.
9. Special dietary requirements or known food allergies.
10. Pregnancy or breastfeeding.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Proteomics and metabolomics changes after diet intervention | 5 weeks
  Changes of plasma, urine, tear proteomics and metabolomics after diet intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No